CLINICAL TRIAL: NCT02639884
Title: Correlation of Endoscopic View of Airway Obstruction With RRa Signal in OSA Patients Under Dexmedetomidine Anesthesia Monitored With SedLine EEG
Brief Title: Correlation Endoscopic View of Airway Obstruction With RRa in OSA Patients Under DEX Monitored With SedLine EEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DROV0007
Record Dates: First submitted 2015-12-11; First posted 2015-12-28 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Evaluation Group (Experimental): All subjects will be enrolled into the evaluation group and will receive SedLine EEG and RRa monitoring
  Interventions: Device: SedLine EEG; Device: RRa monitoring

INTERVENTIONS:
Device: SedLine EEG
Device: RRa monitoring

SUMMARY:
Patients with obstructive sleep apnea (OSA) could have several anatomical causes of obstruction. A sleep endoscopy study is a technique to help determine the anatomical cause of OSA. This study will be using standard of care practice and infuse dexmedetomidine (DEX) to induce sleep. The goals of the study are to (1) confirm airway obstruction with endoscopic view and correlate that with Acoustic Respiratory Rate (RRa) signal at the moment of airway obstruction, and (2) characterize the EEG signals when subjects are under DEX sedation alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients more than 18 years old with American Society of Anesthesiologists (ASA) classification of I, II, or III.
* Patients undergoing sedation for sleep endoscopy with DEX alone, and possible surgical follow-up.

Exclusion Criteria:

* ASA classification higher than III.
* Any deformities or diseases that may prevent application of SedLine (Masimo Sedation Monitoring) or RAM (Masimo Rainbow Acoustic Monitoring) sensors with a proper fit
* Inability to obtain any physiological, vital, demographics and real time anaesthesia data
* Subjects who have known intolerance to any of the drugs to be used according to the study protocol
* Subjects deemed not suitable for study at the discretion of the Principal Investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Drover, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Evaluation Group: All subjects will be enrolled into the evaluation group and will receive SedLine EEG and RRa monitoring
  SedLine EEG
  RRa monitoring
Period: Overall Study
Arm/Group | Evaluation Group
Started | 51
Completed | 47
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Evaluation Group
Number analyzed (Participants) | 47
Age, Continuous [Mean (Full Range); unit: years] | 52 [26 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 35
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects in Which Electroencephalogram (EEG) Signals is Collected
Description: Subjects enrolled into the study will have the SedLine sensor placed on the subject to collect EEG signals.
Time Frame: One visit
Measure: Count of Participants; unit: Participants
Arm/Group | Evaluation Group
Number analyzed (Participants) | 47
Participants | 47

2. Primary Outcome: Number of Subjects in Which Acoustic Respiratory Rate (RRa) Signals is Collected
Description: All subjects enrolled into the study will receive the RAM sensor in order to records RRa signals.
Time Frame: One visit
Measure: Count of Participants; unit: Participants
Arm/Group | Evaluation Group
Number analyzed (Participants) | 47
Participants | 47

ADVERSE EVENTS:
Time Frame: During the data collection period, which could of lasted up to 8 hours.
Arm/Group | Evaluation Group
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT02639884/Prot_SAP_000.pdf